CLINICAL TRIAL: NCT02872961
Title: Relationship Between Small Intestinal Bacterial Overgrowth (SIBO) and Immune System Activation in Childhood Abdominal Pain-Related Functional Gastrointestinal Disorders (FGIDs)
Brief Title: SIBO, Immune Activation, and FGIDs in Children
Acronym: SIBO
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Melissa R Van Arsdall, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-11-0726
Record Dates: First submitted 2016-06-09; First posted 2016-08-19 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Small Intestinal Bacterial Overgrowth; Irritable Bowel Syndrome; Functional Dyspepsia; Functional Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Small intestinal aspirate (fluid) will have bacterial DNA extracted
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SIBO Positive: Positive small bowel aspirate culture and/or positive glucose breath test
- SIBO Negative: Negative small bowel aspirate culture and negative glucose breath test

SUMMARY:
PURPOSE: This study will evaluate the relationships between small intestinal bacterial overgrowth (SIBO), immune activation, inflammation, and symptoms in pediatric abdominal pain-related functional gastrointestinal disorders (FGIDs), i.e., irritable bowel syndrome (IBS), functional dyspepsia (FD), & functional abdominal pain (FAP), to better understand the role of SIBO in their pathogenesis. DESIGN & PROCEDURES: Cross-sectional study. Subjects: Patients followed at the UT-Houston Pediatric GI clinic, aged 4-17 years, undergoing endoscopic evaluation of abdominal pain, meeting Rome III diagnostic criteria for IBS, FD, or FAP, without evidence of an organic etiology of abdominal pain upon routine laboratory, radiologic, endoscopic, histologic evaluation. Sample Size: At least 30 patients, ≥ 15 with SIBO (i.e., positive small bowel aspirate culture and/or glucose breath hydrogen test), and ≥15 without SIBO. Sample Materials: Small bowel biopsies and aspirates, serum, breath samples, symptom questionnaire responses. Measures: 1) Immune activation & inflammation - measured by serum cytokine levels & small intestinal tissue inflammatory cell infiltration & cytokine levels. 2) Symptoms - measured by Abdominal Pain Index, Wong-Baker FACES™ Pain Rating Scale, Questionnaire on Pediatric Gastrointestinal Symptoms - Rome III Version. 3) Small bowel microbiota analysis - assessed by 454 pyrosequencing. RISKS & POTENTIAL BENEFITS: Aside from the risks associated with routine endoscopy with biopsies, which would occur even without study enrollment, the risks associated with serum collection, one extra biopsy specimen collection, small bowel aspirate collection, completion of pain scales/ questionnaires, and the glucose breath hydrogen test for the purposes of the study are minimal. POTENTIAL IMPACT: This study should yield valuable information regarding the relationships between SIBO, immune activation, inflammation, and symptoms in pediatric IBS, FD, and FAP. Potential biomarkers to support the diagnosis of these FGIDs and novel targets for therapy, such as immune molecules and previously unrecognized bacterial phylotypes and species possibly contributing to disease pathogenesis, may be identified. Also, determining the reliability of the glucose breath hydrogen test vs. small bowel aspirate culture in the diagnosis of SIBO in this setting may enable the physician to avoid invasive and costly procedures in the diagnostic work-up of children with these FGIDs.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patient, aged 4-17 years, upon initial evaluation for abdominal pain.
2. Complaints of abdominal pain for at least 2 months upon entry into the study.
3. Esophagogastroduodenoscopy (EGD) ordered by the patient's gastroenterologist for further evaluation / work-up of the patient's abdominal pain.
4. Fulfillment of Rome III criteria for the child/adolescent abdominal pain-related functional gastrointestinal disorders under study (i.e., irritable bowel syndrome, functional dyspepsia, and functional abdominal pain).
5. Signed informed consent for the subject's participation in the study provided by the parent / legal guardian; signed assent signed by study participants 8 years and older.

Exclusion Criteria:

History of short bowel syndrome, defined as clinically significant malabsorption resulting from surgical resection of a substantial portion (≥ 50%) of small intestine, or from complete dysfunction of an extensive portion (≥ 50%) of small bowel. 2. History of other gastrointestinal surgery (except for appendectomy). 3. Other known or suspected motility disorder such as achalasia, gastroparesis, chronic intestinal pseudo-obstruction, dumping syndrome, Hirschprung's disease, or neuromuscular disease.

4. Evidence of enteric infection or infestation on laboratory screening or on mucosal biopsy.

5. Known or suspected of liver, renal, or pancreatic disease. 6. Diabetes mellitus, systemic lupus erythematosus, and/or other systemic disease.

7. Use of antibiotics, mast cell stabilizers, leukotriene modifiers, and/or systemic steroids within 2 weeks preceding the small bowel aspirate culture and biopsies; use of antibiotics or probiotics within 2 weeks of the glucose breath hydrogen test.

8. Use of opiates or benzodiazepines (aside from any given for anesthesia purposes for the endoscopy procedure) or laxatives (aside from any given for bowel preparation for the endoscopy procedure) within 1 week preceding the small bowel aspirate culture and/ or glucose breath hydrogen test.

9. Acute infection or other acute inflammatory process (e.g., upper respiratory tract infection, pneumonia, urinary tract infection, gastroenteritis, pancreatitis, etc.) within the 2 weeks preceding the serum sample and mucosal biopsy collection.

10. Symptomatic from an atopic disorder (i.e., eczema, allergic rhinitis, asthma) within the 2 weeks preceding serum collection for the study.

11. Any evidence of inflammatory bowel disease, celiac disease, H. pylori infection, eosinophilic esophagitis, giardiasis, or other potential organic etiology of abdominal pain upon endoscopic / histologic evaluation.

12. Cancellation of the endoscopy procedure by the subject's gastroenterologist, parent, and/ or legal guardian.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients (ages 4-17 years) presenting to the University of Texas-Houston Pediatric GI Clinic with complaints of abdominal pain and undergoing endoscopy (i.e., esophagogastroduodenoscopy [EGD] and possibly colonoscopy) for further evaluation (at the discretion of the patient's gastroenterologist) will be screened for inclusion into the study at the time that the endoscopic evaluation is ordered by the patient's gastroenterologist.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain Index | Baseline
  To further evaluate symptom severity, on the day of endoscopic evaluation, each subject (or the legal guardian, when appropriate) will be asked to complete the Abdominal Pain Index, which is comprised of five items assessing the frequency, duration, and intensity of abdominal pain episodes the subject has experienced during the previous two weeks. This index was previously validated as a clinical measure of abdominal pain in pediatric patients. Responses to the five pain ratings are standardized, and the Z-scores are averaged to yield an index of abdominal pain.

SECONDARY OUTCOMES:
Duodenal fluid microbiota | Baseline
  Small bowel aspirate specimens of 10 patients from each group (20 total samples) will be randomly selected for further analysis. The tubes will be batched, and the preserved samples will be processed (via microbial DNA extraction, followed by bacterial 16S rRNA gene amplification via PCR), after which deep pyrosequencing analysis of the PCR-amplified 16S rRNA genes will be performed. Pyrosequencing data is processed using the Ribosomal Database Project (RDP) pyrosequencing pipeline (http://pyro.cme.msu.edu/). Statistical differences in the diversity and phylogenetic composition of bacteria in the specimens will be assessed by using the online analysis tools at the RDP pyrosequencing pipeline website and by using both the standard and quantitative UniFrac analyses.
Serum biomarker levels | Baseline
  Levels of key circulating gut biomarkers of inflammation will be measured in serum samples; specifically, levels of IL-1-β, IL-6, IL-8, IL-10, IL-12p70, IFN-γ,TNF-α, and osteoprotegerin), intestinal barrier function (TIMP-1), and GI motility (BDNF) will be measured.
Duodenal tissue inflammatory cell infiltration | Baseline
  Mucosal immune cells from duodenal biopsy specimens will be characterized using Giemsa staining for identification of mast cells and antibodies directed against CD4, CD8 (T-cell markers), and CD20 (B-cell marker) using accepted methods for immunohistochemistry. Quantification of immune cells will be performed on both the hematoxylin and eosin (e.g., total immune cells, lymphocytes, monocytes, eosinophils, basophils) and immunohistochemically stained sections (e.g., mast cells, T-lymphocytes, B-lymphocytes).
Duodenal tissue toll-like receptor expression | Baseline
  Small intestinal toll-like receptor expression will be determined via immunohistochemical staining using established protocols. Levels of the following toll-like receptors will be checked: TLR-2, TLR-4, TLR-5, TLR-9 as these toll-like receptors recognize bacterial ligands and are elevated in inflammatory conditions.
Duodenal tissue cytokine levels | Baseline
  The following cytokine levels will be measured in the small intestinal tissue lysate: Human IL-1-β, IL-6, IL-8, IL-10, IL-12p70, IFN-γ, and TNF-α.
Wong-Baker FACES Pain Rating Scale | Baseline
  To further assess the subject's abdominal pain severity, on the day of endoscopic evaluation, each subject (or the legal guardian, when appropriate) will be asked to rate the subject's current pain, average pain over the preceding two weeks, and worst pain experienced during the preceding two weeks using the Wong-Baker FACES™ Pain Rating Scale. This scale has been validated for use in children and consists of faces showing varying degrees of discomfort, along with corresponding descriptions of the pain and numbers to rate pain.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R Van Arsdall, MD, Principal Investigator — The University of Texas of Health Science Center at Houston
Locations (1):
- The University of Texas of Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided